CLINICAL TRIAL: NCT05355519
Title: Advances in Patient Safety Through Simulation Research
Brief Title: Obstetric Life Support, a Curriculum to Effectively Resuscitate Pregnant Patients Experiencing Cardiac Arrest.
Acronym: OBLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: UConn Health (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrea Shields, Associate Professor of Obstetrics & Gynecology Division of Maternal Fetal Medicine Program Director, Maternal Fetal Medicine Fellowship University of Connecticut School of Medicine, UConn Health
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 22X-137; 5R18HS026169 (AHRQ)
Record Dates: First submitted 2022-04-21; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Cardiac Arrest; Pregnancy Related
Keywords: The Obstetric Life Support Program (OBLS)
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: The investigators will perform a prospective, single-blinded randomized cross-over trial of the OBLS intervention.
Who Masked: Outcomes Assessor
Masking Description: Megacode evaluators will be masked to the arm in which the participants are randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curriculum and Instructor-Led Course (Active Comparator): Participants first complete an online cognitive assessment. Once complete, staff email the electronic curriculum for participants to read. On a specific day, participants will go to the designated center to participate in an instructor-led course and simulated medical scenarios and complete megapode and online cognitive assessment. After a washout period of six months, participants return to the designated center to participate in simulated medical scenarios and complete the online cognitive assessment again. After a second washout period of six months, participants will take the online cognitive assessment again.
  Interventions: Other: Electronic curriculum and instructor-led course, then placebo
- Placebo (Placebo Comparator): On a specific day, participants will go to a designated center to complete an online cognitive assessment and participate in simulated medical scenarios. Once complete, study staff will email the electronic curriculum for participants to read. After a washout period of six months, participants will return to the designated center to participate in an instructor-led course and simulated medical scenarios and complete a megapode and online cognitive assessment. After a second washout period of six months, participants will take an online cognitive assessment again.
  Interventions: Other: Placebo, then electronic curriculum and instructor-led course

INTERVENTIONS:
Other: Electronic curriculum and instructor-led course, then placebo — Electronic curriculum and instructor-led course
  Arms: Curriculum and Instructor-Led Course
Other: Placebo, then electronic curriculum and instructor-led course — Electronic curriculum and instructor-led course
  Arms: Placebo

SUMMARY:
The objective of the study is to determine if Obstetric Life Support Program (OBLS) has an effect on the confidence and skills knowledge in participants.

DETAILED DESCRIPTION:
Enrolled participants with healthcare experience will be randomized to intervention with an electronic curriculum and instructor-led course or placebo first and then will be crossed over to receive the intervention. Participants will undergo assessments pre and post intervention, as well as repeat assessments after three washout periods separated by six months each.

ELIGIBILITY:
Inclusion Criteria:

PH

1. All genders
2. EMS healthcare providers of all levels including basic, advanced, paramedics; firefighters, law enforcement officers, and trainees in any of these programs.
3. 18 years old or older
4. Ability to read, write and speak in English

IH

1. All genders
2. Emergency medicine providers (ED, FP, ICU) surgeons (OB), anesthesiologists, trainees of GME, and nurses from ED, FP, ICU/NICU, or OB/L&D.
3. 18 years or older
4. Ability to read, write and speak in English

Exclusion Criteria:

1. Participants included in the pilot-testing sessions
2. Participants from other medical specialties not listed in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Mean Participant Knowledge Assessment | From baseline to immediately upon completing training
  Mean (standard deviation) of participant knowledge assessment scores post-training stratified by treatment arm. Minimum value is zero and maximum value is 100. A higher score means a better outcome.
Comparison of Scores Between Two Arms | Immediately upon completing training
  Mean (standard deviation) of participant megacode checklist scores post-training stratified by treatment arm.
  Minimum value is zero and maximum value is 200. A higher score means a better outcome.

SECONDARY OUTCOMES:
Self-Reported Confidence Level in Assessing and Managing Critical Care Scenarios in Pregnant Patients | From baseline to 6 months
  Frequency (percent) of participants who self-report that they are confident or very confident in managing procedures in pregnant patients.
Self-Reported Confidence Level in Assessing and Managing Critical Care Scenarios in Pregnant Patients | From baseline to 12 months
  Frequency (%) of participants who self-report that they are confident or very confident in managing procedures in pregnant patients.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Shields, MD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collier AY, Molina RL. Maternal Mortality in the United States: Updates on Trends, Causes, and Solutions. Neoreviews. 2019 Oct;20(10):e561-e574. doi: 10.1542/neo.20-10-e561. PMID 31575778
- [Background] Hameed AB, Lawton ES, McCain CL, Morton CH, Mitchell C, Main EK, Foster E. Pregnancy-related cardiovascular deaths in California: beyond peripartum cardiomyopathy. Am J Obstet Gynecol. 2015 Sep;213(3):379.e1-10. doi: 10.1016/j.ajog.2015.05.008. Epub 2015 May 13. PMID 25979616
- [Background] Briller J, Koch AR, Geller SE; Illinois Department of Public Health Maternal Mortality Review Committee Working Group. Maternal Cardiovascular Mortality in Illinois, 2002-2011. Obstet Gynecol. 2017 May;129(5):819-826. doi: 10.1097/AOG.0000000000001981. PMID 28383382
- [Background] Jeejeebhoy FM, Zelop CM, Lipman S, Carvalho B, Joglar J, Mhyre JM, Katz VL, Lapinsky SE, Einav S, Warnes CA, Page RL, Griffin RE, Jain A, Dainty KN, Arafeh J, Windrim R, Koren G, Callaway CW; American Heart Association Emergency Cardiovascular Care Committee, Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation, Council on Cardiovascular Diseases in the Young, and Council on Clinical Cardiology. Cardiac Arrest in Pregnancy: A Scientific Statement From the American Heart Association. Circulation. 2015 Nov 3;132(18):1747-73. doi: 10.1161/CIR.0000000000000300. Epub 2015 Oct 6. PMID 26443610
- [Background] Goodwin AP, Pearce AJ. The human wedge. A manoeuvre to relieve aortocaval compression during resuscitation in late pregnancy. Anaesthesia. 1992 May;47(5):433-4. doi: 10.1111/j.1365-2044.1992.tb02228.x. PMID 1599071
- [Background] Jeejeebhoy FM, Zelop CM, Windrim R, Carvalho JC, Dorian P, Morrison LJ. Management of cardiac arrest in pregnancy: a systematic review. Resuscitation. 2011 Jul;82(7):801-9. doi: 10.1016/j.resuscitation.2011.01.028. Epub 2011 May 6. PMID 21549495
- [Background] Lipman S, Cohen S, Einav S, Jeejeebhoy F, Mhyre JM, Morrison LJ, Katz V, Tsen LC, Daniels K, Halamek LP, Suresh MS, Arafeh J, Gauthier D, Carvalho JC, Druzin M, Carvalho B; Society for Obstetric Anesthesia and Perinatology. The Society for Obstetric Anesthesia and Perinatology consensus statement on the management of cardiac arrest in pregnancy. Anesth Analg. 2014 May;118(5):1003-16. doi: 10.1213/ANE.0000000000000171. PMID 24781570
- [Background] King SE, Gabbott DA. Maternal cardiac arrest--rarely occurs, rarely researched. Resuscitation. 2011 Jul;82(7):795-6. doi: 10.1016/j.resuscitation.2011.03.029. Epub 2011 Apr 6. No abstract available. PMID 21524838
- [Derived] Shields AD, Vidosh J, Minard C, Thomson B, Annis-Brayne K, Murphy M, Kavanagh L, Roth CK, Lutgendorf MA, Birsner ML, Rahm SJ, Becker LR, Mosesso V, Schaeffer B, Streitz M, Bhalala U, Gresens A, Phelps J, Sutton B, Wagner R, Melvin LM, Zacherl K, Karwoski L, Behme J, Hoeger A, Nielsen PE. Obstetric Life Support Education for Maternal Cardiac Arrest: A Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2445295. doi: 10.1001/jamanetworkopen.2024.45295. PMID 39546311
- See also: Related Info — http://wonder.cdc.gov/ucd-icd10.html
- See also: Related Info — http://apps.who.int/iris/bitstream/handle/10665/194254/9789241565141_eng.pdf;jsessionid=57219BDB4E7FBED75BD83BCDE36F17BF?sequence=1
- See also: Related Info — https://www.unfpa.org/sites/default/files/pub-pdf/9789241507226_eng.pdf